CLINICAL TRIAL: NCT02169336
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Evaluation of the Efficacy, Safety, and Pharmacokinetics of Intranasal Dexmedetomidine for Postoperative Analgesia Following Bunionectomy
Brief Title: Placebo-Controlled Evaluation of Intranasal Dexmedetomidine for Postoperative Analgesia Following Bunionectomy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of observed efficacy
Sponsor: Baudax Bio (Industry)
Collaborators: Lotus Clinical Research, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REC-13-012
Record Dates: First submitted 2014-06-17; First posted 2014-06-23 (Estimated); Results first posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-11

CONDITIONS: Pain, Post-operative
Keywords: Bunion; Bunionectomy; Pain; Analgesia; dexmedetomidine; intranasal
MeSH Terms: conditions — Pain, Postoperative; Bunion; Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- DEX-IN 35mcg (Experimental): DEX-IN 35mcg every 6 hours for 48 hours. DEX-IN 35mcg PRN for up to 3 additional days.
  Interventions: Drug: Intranasal Dexmedetomidine
- DEX-IN 50mcg (Experimental): DEX-IN 50mcg every 6 hours for 48 hours. DEX-IN 50mcg PRN for up to 3 additional days.
  Interventions: Drug: Intranasal Dexmedetomidine
- IN Placebo (Placebo Comparator): IN Placebo every 6 hours for 48 hours. IN Placebo PRN for up to 3 additional days.
  Interventions: Other: Intranasal Placebo

INTERVENTIONS:
Drug: Intranasal Dexmedetomidine
  Arms: DEX-IN 35mcg; DEX-IN 50mcg
Other: Intranasal Placebo
  Arms: IN Placebo

SUMMARY:
The primary objective of this study is to evaluate the analgesic efficacy of two dose levels of DEX-IN compared with placebo, using the summed pain intensity difference over the first 48 hours (SPID48) in subjects with acute moderate to severe pain following unilateral bunionectomy.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily provide written informed consent.
* Male or female between 18 and 70 years of age, inclusive.
* Be scheduled to undergo a primary unilateral first metatarsal bunionectomy repair
* Be American Society of Anesthesiology (ASA) physical class 1 or 2.
* Female subject are eligible only if all the following apply:

  * Not pregnant;
  * Not lactating;
  * Not planning to become pregnant during the study;
  * Be surgically sterile; or at least two year post menopausal; or have a monogamous partner who is surgically sterile; or is practicing double-barrier contraception; or practicing abstinence; or using an insertable, injectable, transdermal, or combination oral contraceptive.
* Male subjects must be surgically sterile or commit to the use of a reliable method of birth control
* Have a body mass index ≤35 kg/m2
* Be able to understand the study procedures, comply with all study procedures, and agree to participate in the study program.

Exclusion Criteria:

* Have a known allergy to dexmedetomidine or any excipient DEX-IN/placebo or to any peri- or postoperative medications used in this study.
* Have a clinically significant abnormal clinical laboratory tests value.
* Have history of or positive test results for HIV, or hepatitis B or C.
* Have a history or clinical manifestations of significant renal, hepatic, cardiovascular, metabolic, neurologic, psychiatric, or other condition that would preclude participation in the study.
* Have a history of migraine or frequent headaches, seizures, or are currently taking anticonvulsants.
* Have another painful physical condition that may confound the assessments of post operative pain.
* Have a history of syncope or other syncopal attacks.
* Have evidence of a clinically significant 12 lead ECG abnormality.
* Have a history of alcohol abuse (regularly drinks > 4 units of alcohol per day; 8 oz. beer, 3 oz. wine, 1 oz. spirits) or prescription/illicit drug abuse..
* Have positive results on the urine drug screen or alcohol breath test indicative of illicit drug or alcohol abuse.
* Have a history or evidence of orthostatic hypotension.
* Have a resting heart rate of <50 beats per minutes or systolic blood pressure <100mmHg.
* Have been receiving or have received chronic opioid therapy defined as greater than 15 morphine equivalents units per day for greater than 3 out of 7 days per week over a one-month period within 12 months.
* Use concurrent therapy that could interfere with the evaluation of efficacy or safety, such as any drugs which in the investigator's opinion may exert significant analgesic properties or act synergistically with DEX-IN.
* Unable to discontinue medications, that have not been at a stable dose for at least 14 days prior to the scheduled bunionectomy procedure, within 5 half lives of the specific prior medication (or, if half life is not known, within 48 hours) before dosing.
* Have utilized any intranasal medications within the preceding 10 days.
* Have signs or a history of significant rhinitis or rhinorrhea (constant or chronic), nasal polyps, mucosal lesions of the nostril, postnasal drip of any etiology (constant or chronic), nasal ulcers, septal perforation or deviation, any nasal surgery, anosmia, nasal piercings, or frequent nosebleeds or other nasal pathology, that is sufficient to interfere with IN drug delivery.
* Have had an upper respiratory tract infection within 14 days of screening.
* Have utilized corticosteroids, either systemically, inhalational either intranasally or oral, or by intra-articular injection, within 14 days prior to the study.
* Have received any investigational product within 30 days before dosing with study medication.
* Have previously received DEX-IN in clinical trials, or had bunionectomy in the last 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Singla, MD, Principal Investigator — Lotus Clinical Research, LLC
Locations (3):
- United States (3):
  - Trovare Clinical Research, Inc., Bakersfield, California
  - Lotus Clinical Research, LLC, Pasadena, California
  - Endeavor Clinical Trials, P.A., San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- DEX-IN 35mcg: DEX-IN 35mcg every 6 hours for 48 hours. DEX-IN 35mcg PRN for up to 3 additional days.
  Intranasal Dexmedetomidine
- DEX-IN 50mcg: DEX-IN 50mcg every 6 hours for 48 hours. DEX-IN 50mcg PRN for up to 3 additional days.
  Intranasal Dexmedetomidine
- IN Placebo: IN Placebo every 6 hours for 48 hours. IN Placebo PRN for up to 3 additional days.
  Intranasal Placebo
Period: Overall Study
Arm/Group | DEX-IN 35mcg | DEX-IN 50mcg | IN Placebo
Started | 31 | 32 | 32
Completed | 27 | 28 | 29
Not Completed | 4 | 4 | 3
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Adverse Event | 2 | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Subject declined to continue dosing | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DEX-IN 35mcg | DEX-IN 50mcg | IN Placebo | Total
Number analyzed (Participants) | 31 | 32 | 32 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (14.53) | 44.6 (12.21) | 44.6 (13.93) | 44.2 (13.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 28 | 27 | 78
  Male | 8 | 4 | 5 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 10 | 14 | 38
  Not Hispanic or Latino | 17 | 22 | 18 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 8 | 11 | 24
  White | 24 | 24 | 21 | 69
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Summed Pain Intensity Difference Over the First 48 Hours (SPID48).
Description: Pain intensity was recorded using a Numeric Rating Scale (Range 0-10) where 0 equates to no pain, and 10 equates to the worst pain imaginable. Pain intensity scores were to be recorded at the following time points: 0.25, 0.5, 0.75, 1, 2, 4, and 6 hours post Dose 1. Thereafter pain assessments were to be recorded every 2 hours until 48 hours. Pain intensity differences from baseline at each time point were calculated and a time weighted SPID was then calculated. Time weighted SPID calculations were computed by multiplying a weight factor to each score prior to summation. The weight factor at each time point was the time elapsed since the previous observation.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DEX-IN 35mcg | DEX-IN 50mcg | IN Placebo
Number analyzed (Participants) | 31 | 32 | 32
units on a scale | 36.871 (93.7979) | 44.719 (79.0590) | 51.227 (100.3288)

ADVERSE EVENTS:
Time Frame: All AEs were to be recorded beginning after administration of study medication through the final follow-up assessment. In addition, if the investigator became aware of the occurrence of a SAE within 30 days of the last visit, the SAE was to be reported.
Arm/Group | DEX-IN 35mcg | DEX-IN 50mcg | IN Placebo
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 28/31 | 30/32 | 26/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DEX-IN 35mcg (N=31) | DEX-IN 50mcg (N=32) | IN Placebo (N=32)
Constipation (Gastrointestinal disorders) | 2 | 2 | 1
Nausea (Gastrointestinal disorders) | 11 | 8 | 14
Vomiting (Gastrointestinal disorders) | 4 | 3 | 6
Fatigue (General disorders) | 7 | 6 | 8
Blood Pressure Decreased (Investigations) | 4 | 6 | 0
Disturbance in Attention (Nervous system disorders) | 5 | 4 | 5
Dizziness (Nervous system disorders) | 6 | 3 | 5
Headache (Nervous system disorders) | 5 | 2 | 6
Somnolence (Nervous system disorders) | 20 | 17 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Nasal Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 4
Hypotension (Vascular disorders) | 1 | 3 | 0

LIMITATIONS AND CAVEATS:
An interim analysis was performed that focused on the primary efficacy endpoint (SPID48). Observed effect size was determined for purposes of final sample size determination. The study was terminated following the interim analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Discussion and/or publication of data generated is not permitted without the prior written consent of the sponsor.